CLINICAL TRIAL: NCT02155010
Title: Hemodynamic Effect of Dexmedetomidine on Heavy Bupivacaine Spinal Anesthesia
Brief Title: Dexmedetomidine in Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2014-003
Record Dates: First submitted 2014-05-22; First posted 2014-06-04 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Blood Pressure; Anxiety
Keywords: Dexmedetomidine; Spinal anesthesia
MeSH Terms: conditions — Anxiety Disorders | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): IV dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine with heavy bupivacaine (Active Comparator): IV dexmedetomidine infusion after intrathecal injection of heavy bupivacaine
  Interventions: Drug: Dexmedetomidine with heavy bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Dexmedetomidine with heavy bupivacaine — Dexmedetomidine infusion after IT of heavy bupivacaine
  Other Names: Precedex; Marcaine
  Arms: Dexmedetomidine with heavy bupivacaine

SUMMARY:
Patients were randomized into two groups, A group and B group. A group and B group patients are injected intravenous dexmedetomidine after intrathecal injection (IT) of heavy bupivacaine and injected intravenous dexmedetomidine before IT of heavy bupivacaine, respectively.

The investigators will compare of hemodynamics and patient's comfortability between two groups.

DETAILED DESCRIPTION:
A and B group patients will intravenous inject dexmedetomidine 1mcg/kg for 10 minute loading infusion and 0.2mcg/kg/hr for continuous infusion. A group receive intravenous dexmedetomidine after procedure, and B group receive intravenous dexmedetomidine before procedure. Both group patients will hydrate 6 ml/kg crystalloid solution and will evaluated patient's anxiety and comfortability perioperative period. Vital signs will record 5 minutes interval at operating room and post-anesthetic care units.

ELIGIBILITY:
Inclusion Criteria:

* 20 - 60 aged patients
* orthopedic operation undergoing spinal anesthesia

Exclusion Criteria:

* more than American society of anesthesiologists classification 3
* hypertension
* diabetes mellitus
* heart disease (bradycardia, atrioventricular block)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hwa Lee, MD, Principal Investigator — Inje University Haeundae Paik Hospital
Locations (1):
- Inje University, Haeundae paik hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 3 years of study completion.

REFERENCES:
- [Derived] Kang E, Lee KH, Jeon SY, Lee KW, Ko MJ, Kim H, Kim YH, Jung JW. The timing of administration of intravenous dexmedetomidine during lower limb surgery: a randomized controlled trial. BMC Anesthesiol. 2016 Nov 21;16(1):116. doi: 10.1186/s12871-016-0282-2. PMID 27871236

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine Before Bupivacaine: IV dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
  Dexmedetomidine: Dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
- Dexmedetomidine After Bupivacaine: IV dexmedetomidine infusion after intrathecal injection of heavy bupivacaine
  Dexmedetomidine with heavy bupivacaine: Dexmedetomidine infusion after IT of heavy bupivacaine
Period: Overall Study
Arm/Group | Dexmedetomidine Before Bupivacaine | Dexmedetomidine After Bupivacaine
Started | 37 | 37
Completed | 31 | 31
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Before Spinal Anesthesia: IV dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
  Dexmedetomidine: Dexmedetomidine infusion before intrathecal injection of heavy bupivacaine
- After Spinal Anesthesia: IV dexmedetomidine infusion after intrathecal injection of heavy bupivacaine
  Dexmedetomidine with heavy bupivacaine: Dexmedetomidine infusion after IT of heavy bupivacaine
- Total: Total of all reporting groups
Arm/Group | Before Spinal Anesthesia | After Spinal Anesthesia | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.74 (12.27) | 35.87 (11.22) | 37.31 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 15 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypotension
Description: We compare incidence rate of hypotension during infusion of dexmedetomidine
Time Frame: up to 3 hours
Measure: Number; unit: participants
Arm/Group | Before Spinal Anesthesia | After Spinal Anesthesia
Number analyzed (Participants) | 31 | 31
participants | 15 | 5

2. Secondary Outcome: Patient's Anxiety
Description: We compared patient's anxiety using spielberger's state-trait anxiety inventory before and after surgery. This consists of two self-evaluation scales designed to assess state-anxiety and trait-anxiety. Each scale contains 20 items, each of which is rated from 1 to 4. Clinically significant levels of state or trait-anxiety were defined as scores >50 on the state- or trait-anxiety scale. State or trait-anxiety inventory's minimal score is 20 and maximal score is 80. We analyzed State Anxiety Inventory scale before and after surgery.
Time Frame: up to 3 days
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Before Spinal Anesthesia | After Spinal Anesthesia
Number analyzed (Participants) | 31 | 31
points
  State Anxiety Inventory (Preoperative) | 43.65 (14.24) | 45.52 (12.01)
  State Anxiety Inventory (discharge from PACU) | 37.03 (10.51) | 38.55 (8.04)
  State Anxiety Inventory (postoperative first day) | 34.90 (9.03) | 34.55 (8.64)

ADVERSE EVENTS:
Time Frame: <24 hours
Arm/Group | Before Spinal Anesthesia | After Spinal Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
We did not assess the differences among the groups regarding postoperative analgesic consumption and the duration of sensory or motor bloakade produced by spinal anesthesia with dexmedetomidine infusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No